CLINICAL TRIAL: NCT03876522
Title: Prospective, Longitudinal, Observational Study of the Natural History and Functional Status of Patients With Lafora Disease
Brief Title: Natural History and Functional Status Study of Patients With Lafora Disease
Status: Completed | Type: Observational
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAF-NHS
Record Dates: First submitted 2019-01-10; First posted 2019-03-15 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Lafora Disease
Keywords: Lafora Disease; EPM2A; EPM2B; Myoclonus epilepsy; Myoclonic seizures; Glycogen storage disease
MeSH Terms: conditions — Lafora Disease; Epilepsies, Myoclonic; Seizures; Glycogen Storage Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected and used for evaluations of potential biomarkers of Lafora disease progression.
  Cerebral spinal fluid (CSF) samples will be collected and used for safety evaluations and assessments of potential biomarkers of Lafora disease progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lafora Disease Patients: Documented genetic diagnosis of Lafora disease; clinical diagnosis of Lafora disease and a sibling with a known mutation in EPM2A or EPM2B; clinical diagnosis of Lafora disease and a previously undescribed mutation in EPM2A or EPM2B; asymptomatic siblings if mutation positive prior to enrollment.

SUMMARY:
A natural history and functional status study to characterize the clinical disease course in Lafora disease patients using standardized, quantitative evaluations and to identify useful biomarkers and clinical outcome measures for use in future Lafora treatment studies.

ELIGIBILITY:
Inclusion Criteria:

1. Documented genetic diagnosis of Lafora disease based on mutations in both alleles of either the EPM2A or the EPM2B gene and a sibling with a known mutation in EPM2A or EPM2B.
2. Able and willing to comply with the study protocol, including travel to Study Center, procedures, measurements and visits, including:

   1. Adequately supportive psychosocial circumstances, in the opinion of the Investigator
   2. Caregiver/trial partner committed to facilitate patient's involvement in the study who is reliable, competent, at least 18 years of age.
   3. Adequate visual and auditory acuity for neuropsychological testing

Exclusion Criteria:

1. Any known genetic abnormality, including chromosomal aberrations that confound the clinical phenotype
2. Subjects with:

   1. complete absence of speech OR
   2. inability to perform any activities of daily living OR
   3. who are completely bedridden.
3. Current participation in an interventional or therapeutic study
4. Receiving an investigational drug within 90 days of the Baseline Visit
5. Prior or current treatment with gene or stem cell therapy
6. Any other diseases which may significantly interfere with the assessment of Lafora disease.
7. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Global Lafora patient population
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Changes over time in symptom-directed physical exams, measured by height assessment | 24 Months
Changes over time in symptom-directed physical exams, measured by weight assessment | 24 Months
Changes over time in symptom-directed physical exams, measured by head, eyes, ears, nose, and throat assessment (HEENT) | 24 Months
Changes over time in symptom-directed physical exams, measured by cardiovascular assessment | 24 Months
Changes over time in symptom-directed physical exams, measured by musculoskeletal assessment | 24 Months
Changes over time in symptom-directed physical exams, measured by respiratory assessment | 24 Months
Changes over time in symptom-directed physical exams, measured by abdomen assessment | 24 Months
Changes over time in symptom-directed physical exams, measured by skin findings | 24 Months
Changes in disease-related symptoms over time assessed by the Lafora Disease Performance Scale | 24 Months
Seizure frequency, (by type and severity) as recorded in seizure diary | 24 Months
Seizure duration, as measured by awake video EEG | 24 Months
  EEG measured by background activity awake presence of slow waves
Seizure duration, as measured by sleep video EEG | 24 Months
  EEG measured by background activity sleep presence of vertex waves
Change in disease severity using the Lafora Disease Clinical Performance Scale | 24 Months
Change in use of anti-epileptic rescue medication as recorded in seizure diary | 24 Months
Intelligence, as measured by the Leiter International Performance Scale | 24 Months
Cognitive Function, as measured by Woodcock-Johnson IV Tests of Oral Language | 24 Months
Cognitive Function, as measured by Rey Complex Figure Test | 24 Months
Cognitive Function, as measured by Children's Orientation and Amnesia Test (COAT) | 24 Months
Cognitive Function, as measured by Beery Buktenica Developmental Test of Visual Motor Integration | 24 Months
Cognitive Function, as measured by Children's Color Trails Test | 24 Months
Motor function, as measured by Gait Analysis | 24 Months
Caregiver Ratings, as measured by Vineland-II and Burden Scale of Family Caregivers (short form) | 24 Months
Disability, as rated by Pediatric Evaluation of Disability Inventory (PEDI) | 24 Months
Ataxia, as measured by the Scale of Assessment and Rating of Ataxia (SARA) | 24 Months
Motor function, as measured by Six-Minute Walk Test (6MWT) | 24 Months
Motor function, as measured by Timed Up and Go Test (TUG) in ambulatory patients | 24 Months
Motor function, as measured by 9 Hole Pegboard Test | 24 Months
Quality of Life (QoL), as measured by QoL in Epilepsy for Adolescents (QOLIE-AD-48) by age at Screening | 24 Months
Quality of Life (QoL), as measured by QoL in Epilepsy (QOLIE-31P) by age at Screening | 24 Months
Quality of Life (QoL), as measured by QoL in Childhood Epilepsy (QOLCE-55) by age at Screening | 24 Months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - IONIS Investigative Site, Los Angeles, California
  - IONIS Investigative Site, Dallas, Texas
- IONIS Investigative Site, Bologna, Italy
- IONIS Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No